CLINICAL TRIAL: NCT07205406
Title: Effect of Parenting Training on Quality of Life and Parenting in Parents Who Have Children With Intellectual Disabilities
Brief Title: Parenting Training Effect on Quality of Life and Parenting in Parents Who Have Children With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: STIKes Satria Bhakti Nganjuk (Other)
Responsible Party: Principal Investigator, Rahayu Budi Utami, Principal investigator, STIKes Satria Bhakti Nganjuk
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STIKesNganjuk
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Intellectual Disabilities (F70-F79); Quality of Life; Parenting Intervention
Keywords: intellectual disabilities; parenting; quality of life; parenting training
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parenting training group (Experimental): mothers who have children with intellectual disabilities received parenting training in a group for approximately three hours, once a week for 5 weeks. They also received a parenting guidebook for children with intellectual disabilities
  Interventions: Behavioral: group based-parenting training
- control group (No Intervention): mothers who have children with intellectual disabilities received a parenting guidebook for children with intellectual disabilities

INTERVENTIONS:
Behavioral: group based-parenting training — The group received approximately three hours of parenting training once a week for 5 weeks that focused on understanding children with ID in the first week, practical parenting skills in the second week, and how to provide emotional support and regulate parental emotions in the third week. Knowledge and skills were reinforced in the fourth and fifth weeks. The intervention group received training in small groups, each consisting of only 10 participants. The training involved experts in mental health counseling, pediatric nurses, special school teachers, and a motivator.
  Arms: parenting training group

SUMMARY:
We conducted a non-randomized control trial. One hundred and forty-one participants in eleven special schools were included in an intervention group (N=71) to participate in parenteral training once a week for five weeks, and in a control group (N=70). Quality of care was evaluated using the Parenting Sense of Competence (PSOC), and quality of life was evaluated using the World Health Organization Quality of Life (WHOQOL-BREF) before and one week after the intervention. The study used within-group analysis (Wilcoxon test) and intergroup analysis (Mann-Whitney U test) to evaluate the effects of group-based parenting training. The Point-biserial correlation test was used to evaluate the effect size.

DETAILED DESCRIPTION:
This study used a quasi-experimental design, which was conducted based on a pretest-posttest control group. One hundred and forty-one mothers who have children with intellectual disabilities attending special schools in East Java, Indonesia, were recruited and divided into intervention (N=71) and control group (N = 70) according to a special school using a convenience sampling method.

The inclusion criteria were

* having a child aged 7-18 years who has mild and moderate intellectual disabilities
* living in the same house as a child with intellectual disabilities,
* being able to communicate fluently The exclusion criteria were
* having disabilities
* having a child with intellectual disabilities who has a chronic disease
* having a child with intellectual disabilities and other disabilities Parenting quality was evaluated using the Parenting Sense of Competence (PSOC) developed by Gibaud-Wallston and Wandersman, adapted from Johnston and Marsh. Quality of life was evaluated using the World Health Organization Quality of Life (WHOQOL-BREF) (Cronbach Alpha= 0.66-0.8) developed by the WHO . The control and intervention groups were given a parenting guidebook for children with intellectual disabilities. The intervention group received approximately three hours of parenting training once a week for 5 weeks. The intervention group received parenting training focused on understanding children with intellectual disabilities in the first week, practical parenting skills in the second week, and how to provide emotional support and regulate parental emotions in the third week. Knowledge and skills were reinforced in the fourth and fifth weeks. The intervention group received training in small groups, each consisting of only 10 participants. The training involved experts in mental health counseling, pediatric nurses, special school teachers, and a motivator. The Wilcoxon and Mann-Whitney U tests were used for continuous variables with non-normal distributions, as well as the Chi-squared test for qualitative variables. The Wilcoxon and Mann-Whitney U tests were used for continuous variables with non-normal distributions. A p-value of less than 0.05 was considered statistically significant. The point-biserial correlation test was used to evaluate the effect size.

ELIGIBILITY:
Inclusion Criteria:

* having a child aged 7-18 years who has mild and moderate intellectual disabilities
* living in the same house as a child with intellectual disabilities
* being able to communicate fluently

Exclusion Criteria:

* having disabilities
* having a child with intellectual disabilities who has a chronic disease
* having a child with intellectual disabilities and other disabilities bilities

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — mothers who have children with intellectual disabilities
Enrollment: 141 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
quality of life of parents who have intellectual diasabilities | 1 week after intervention
  Quality of life of parents was evaluated using the World Health Organization Quality of Life (WHOQOL-BREF) developed by the WHO The WHOQOL-BREF consists of four domains (physical health, psychological, social relationships, and environment) with 26 questions. The total score for each domain is transformed to a scale of 0-100 according to the scoring guidelines.
Parenting quality | 1 week after intervention
  Parenting quality was evaluated using the Parenting Sense of Competence (PSOC) developed by Gibaud-Wallston and Wandersman, adapted from Johnston and Marsh. The PSOC consists of the domains of satisfaction and self-efficacy with parenting, which are assessed with 16 questions, with a satisfaction score ranging from 9 to 54 and a self-efficacy score from 7 to 42.

CONTACTS AND LOCATIONS:
Overall Officials: Rahayu B Utami, Magister, Principal Investigator — STIKes Satria Bhakti Nganjuk
Locations (1):
- Special school, Nganjuk, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenaro C, Flores N, Gutierrez-Bermejo B, Vega V, Perez C, Cruz M. Parental Stress and Family Quality of Life: Surveying Family Members of Persons with Intellectual Disabilities. Int J Environ Res Public Health. 2020 Dec 3;17(23):9007. doi: 10.3390/ijerph17239007. PMID 33287284
- [Background] Grenier-Martin, J., Rivard, M., Patel, S., Lanovaz, M. J., & Lefebvre, C. (2022). Randomized controlled trial on an online training to support caregivers of young children with intellectual and developmental disability managing problem behaviors at home. Journal of Child and Family Studies, 31(12), 3485-3497.
- [Background] Coren E, Ramsbotham K, Gschwandtner M. Parent training interventions for parents with intellectual disability. Cochrane Database Syst Rev. 2018 Jul 13;7(7):CD007987. doi: 10.1002/14651858.CD007987.pub3. PMID 30004571
- [Background] Barratt M, Lewis P, Duckworth N, Jojo N, Malecka V, Tomsone S, Rituma D, Wilson NJ. Parental Experiences of Quality of Life When Caring for Their Children With Intellectual Disability: A Meta-Aggregation Systematic Review. J Appl Res Intellect Disabil. 2025 Jan;38(1):e70005. doi: 10.1111/jar.70005. PMID 39763193
- [Background] Alghamdi SA, Assiri MI, Fallatah RA, Albeladi FM, Alabdulaziz H, Alsaggaf F. Health-promoting activities among Saudi Arabian parents of children with disabilities: A cross-sectional study. Belitung Nurs J. 2025 Jan 26;11(1):75-82. doi: 10.33546/bnj.3624. eCollection 2025. PMID 39877218

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT07205406/Prot_SAP_000.pdf